CLINICAL TRIAL: NCT03335202
Title: Longitudinal Analysis of Respiratory and Intestinal Microbiome in Cystic Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Kiel (Other)
Responsible Party: Principal Investigator, Ingrid Bobis, Dr. med., Oberärztin für Pneumologie, Head of Adult CF Centre UKSH Kiel, Klinik für Innere Medizin I UKSH Kiel, University of Kiel
Other Study IDs: B495/16
Record Dates: First submitted 2017-09-28; First posted 2017-11-07 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Cystic Fibrosis
Keywords: respiratory and intestinal microbiome; antibiotic therapy; cftr modifier; diversity
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Sputum, throat swab and stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- cf patients at the cf centre Kiel: microbiome of cf patients at the cf centre Kiel will be analyzed and correlated to standard cf care.
  Interventions: Diagnostic Test: analysis of microbiome

INTERVENTIONS:
Diagnostic Test: analysis of microbiome — microbial profiling by next generation sequencing

SUMMARY:
Respiratory und intestinal microbiome will bei analyzed during a period of 6 months. In a retrospective analysis it will be looked for correlations between microbiome and cf therapy (e.g. inhaled and systemic antibiotics, cftr modifiers, proton pump Inhibitors, enzymes, nutritional habits), clinical status and self reported outcome.

DETAILED DESCRIPTION:
DNA will be isolated from sputum, throat swabs and stool samples and used for the generation of microbial profiles. Both bacterial and fungal profiles will be analyzed by next generation sequencing.

Clinical outcome parameters (lung function test, weight, calprotectin, elastase, blood parameters, self reported outcome) will be recorded and analyzed along with medication.

ELIGIBILITY:
Inclusion Criteria:

* subject has confirmed diagnosis of cystic fibrosis (sweat chloride >60mmol/l and/or 2 mutations in the cftr gene known to cause cystic fibrosis)
* subject is able to perform informed consent

Exclusion Criteria:

* inability to give informed consent
* antibiotic therapy in the last 4 weeks prior to study start (exception: long term azithromycin therapy, long term antistaphylococcal therapy, long term inhaled antibiotics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult cf patients treated in Adult Cystic Fibrosis Center, Klinik für Innere Medizin I, UKSH Kiel
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2017-09-28 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
respiratory microbiome | 24 weeks
  abundance [operational taxonomic units]
intestinal microbiome | 24 weeks
  abundance [operational taxonomic units]

SECONDARY OUTCOMES:
Forced Exspiratory Volume FEV1 [%pred] | 24 weeks
  performed by bodyplethmograph
weight (kg) | 24 weeks
  for children, height (cm) is also recorded
Quality of life [score] | 24 weeks
  Cystic Fibrosis Questionnaire Revised CFQ-R [score 0-100, higher scores indicating better Quality of Life]
Quality of life [score] | 24 weeks
  Kiel Questionnaire Kiel-Q [score 0-100, higher scores indicating hetter Quality of Life]

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid CF Bobis, MD, Principal Investigator — Klinik für Innere Medizin I, UKSH Kiel
Locations (1):
- Klinik für Innere Medizin I, UKSH KIel, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-09-28): https://cdn.clinicaltrials.gov/large-docs/02/NCT03335202/Prot_000.pdf